CLINICAL TRIAL: NCT00762866
Title: Psychiatric Genotype/Phenotype Project
Brief Title: Psychiatric Genotype/Phenotype Project Repository
Acronym: PGPP
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephan Heckers, Chair of the Department of Psychiatry, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 080606
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders
Keywords: Major Depressive Disorder; Depression; Bipolar I Disorder; Bipolar II Disorder; Bipolar Disorder NOS; Psychotic Disorder; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders; Depression; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Blood, urine, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MDD: Unipolar Major Depressive Disorder, any subtype
- Bipolar: Bipolar I or II Disorder or Bipolar Disorder NOS
- Psychosis: Psychotic Disorder including Schizophrenia, Schizoaffective, Schizophreniform, Brief Psychotic Disorder, and Psychotic Disorder NOS

SUMMARY:
The purpose of this project is to obtain DNA, brain imaging data, other biological samples (e.g., urine, serum), and a comprehensive clinical assessment on patients with schizophrenia and other psychotic disorders, bipolar disorder, major depression, and normal volunteer controls. Understanding the physical and genetic factors related to these disorders will help us make progress in fitting treatments to an individual's needs. Participants will take part in a detailed clinical assessment, two blood draws, and an MRI scan over two visits. Participants will also be asked to provide urine and saliva samples.

DETAILED DESCRIPTION:
The links between psychiatric symptoms and underlying biological processes remain unclear at this time. Unipolar Major Depressive Disorder, Bipolar Disorder, and Schizophrenia are associated with major disruptions in functioning and quality of life. Understanding the causal physiological and genetic factors involved in each of these disorders would allow us to make great strides in tailoring treatment to the individual's needs. Because the etiology of these disorders are likely multifactorial in nature, a study examining a wide range of variables might best allow us to examine the interactions between different factors and to get a better sense of how genes and the brain interact to produce psychiatric disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 16 and 65
2. Able and willing to provide informed consent
3. Able to read and speak English sufficiently to provide consent and answer questions
4. Diagnosis of one of the following:

   * Unipolar Major Depressive Disorder of any subtype
   * Bipolar I, Bipolar II Disorder, or Bipolar Disorder NOS
   * Axis I Psychotic Disorder, which can include the diagnoses of Schizophrenia, Schizoaffective Disorder, Major Depression or Mania with Psychotic Features, Schizophreniform Disorder, Brief Psychotic Episode, or Psychotic Disorder NOS
   * Normal volunteer controls, individuals with no personal history of any Axis I disorder.

Exclusion Criteria:

1. Reported pregnancy or breastfeeding
2. Dementia or delirium
3. Any medical condition that would interfere with participation in the study. This would include, but not be limited to:

   * uncontrolled diabetes, hypothyroidism, Cushing's disease, or other significant endocrine condition (treated endocrine condition is allowed)
   * demyelinating disease
   * HIV infection
   * active hepatitis
   * CNS infection
   * clinically significant and unstable cardiovascular disease
   * any cancer involving the CNS (including metastatic disease)
4. Exclusion criteria for normal control subjects include any history of mental illness or psychotropic drug abuse.
5. Participants will be excluded from the imaging portion of the study if they have any condition deemed to interfere with PET or MRI scanning, such as but not restricted to extreme obesity, metal fragments in eyes, metal implants in the head, or cochlear implant. These participants may still take part in the portion of the study involving the clinical assessment and providing biological samples.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient Mental Health Clinic, Inpatient Psychiatric Hospital, Research Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Brain volume | 2 years
  Observational neuromaging study

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Heckers, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States